CLINICAL TRIAL: NCT05390073
Title: Assessment of Growth Hormone and Insulin-like Growth Factor 1 in Children With Epidermolysis Bullosa Dystrophia
Brief Title: Growth Hormone in EB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Other Study IDs: Growth in EB
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: growth hormone level and insulin like growth factor 1 — laboratory test

SUMMARY:
Growth is extremely affected in epidermolysis bullosa patients

DETAILED DESCRIPTION:
Studying the role of growth hormone and ILGF-1 in EB may pave the to new therapeutic modality that could improve the growth in those children and avoid the irreversible sequelae that affected subjects experience after adulthood

ELIGIBILITY:
Inclusion Criteria:

- Children with EB dystrophica

Exclusion Criteria:

* Adults with the same disease

Ages: 1 Month to 12 Years | Sex: All
Age Groups: Child
Study Population: Children with EB dystrophica
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
level of growth hormone and insulin like growth factor 1 | 2 weeks
  laboratory test

REFERENCES:
- [Derived] El Darouti M, Zaki IS, Mousa N, El Sayed H. Assessment of Growth Hormone and Insulin-Like Growth Factor 1 in Children With Epidermolysis Bullosa Dystrophica. Pediatr Dermatol. 2025 Nov 24. doi: 10.1111/pde.70113. Online ahead of print. PMID 41287410